CLINICAL TRIAL: NCT03991676
Title: Clarifying the Role of Values in Weight Control: A Pilot Study of a Values-Based Intervention to Promote Weight Loss
Brief Title: A Study of a Values-Based Intervention to Promote Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Diane Dallal, Graduate Student, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DrexelUniversity
Record Dates: First submitted 2019-05-19; First posted 2019-06-19 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Behavioral treatment; Values; Values-based behavior change; Autonomous motivation; Acceptance and Commitment Therapy
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: All participants are enrolled into a single condition, consisting of a series of three, once-weekly values-infused weight loss workshops.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Values-Based Behavioral Treatment (Experimental)
  Interventions: Behavioral: Values-Based Behavioral Treatment

INTERVENTIONS:
Behavioral: Values-Based Behavioral Treatment — The values-based behavioral treatment will consist of a series of three, once-weekly weight loss workshops infused with techniques to elicit values clarification and awareness in moments of dietary decision-making, and to enhance autonomous motivation for behavior change.

SUMMARY:
More than 160 million American adults are overweight or obese. Existing weight loss interventions from self-help to gold standard behavioral treatments, while often effective, do not sufficiently maintain motivation to adhere to dietary goals in the face of powerful biological and environmental influences to consume highly palatable foods. Clarification and awareness of values, a staple of acceptance-based treatments drawn from Acceptance and Commitment Therapy, are thought to enhance autonomous motivation to engage in behaviors consistent with one's personal life values (e.g., health) in the presence of countervailing forces (e.g., hunger, deprivation). However, the independent efficacy of values clarification and awareness in facilitating weight control has never been tested. This pilot study seeks to investigate the feasibility and acceptability of a series of three weight loss workshops (based off the gold standard) infused with values clarification and awareness techniques to promote weight control. Participants will be asked to follow a reduced-calorie dietary prescription while holding their values in mind in moments of dietary decision-making over the course of one month. The primary aims of this study are to: 1) develop the series of values-infused workshops, using participant feedback to iterate and improve the treatment manual; and 2) evaluate treatment acceptability. Secondary aims are: 1) to evaluate whether clinically meaningful changes in measures of values clarification and values awareness occur; 2) to evaluate whether the intervention will lead participants to experience clinically meaningful changes in values-congruent weight control behaviors; 3) to evaluate whether the intervention will lead participants to experience clinically meaningful changes in weight; and 4) to evaluate theorized mechanisms of action in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25-55 kg/m2
* 18-70 years of age
* Have a desire to lose weight
* Own a smartphone
* Live in the Philadelphia area
* Provide informed consent

Exclusion Criteria:

* Any medical or psychiatric conditions (e.g., eating disorder, diabetes) that may pose a risk to the participant during the intervention, cause a change in weight or appetite, or interfere with ability to adhere to diet recommendations
* Recent change in medication dosage that could affect weight or appetite
* Current or planned pregnancy in the next month
* Planned move out of the Philadelphia area in the next month
* History of bariatric surgery
* Weight loss of ≥5% in the last six months
* Concurrent behavioral therapy targeting weight control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Participant acceptability and satisfaction with the intervention | Measured at post-treatment (1 month).
  Participant acceptability and satisfaction with the intervention will be assessed using an idiosyncratic self-report Acceptability Questionnaire, developed for the present study. Questions include items assessing how satisfied participants were with the intervention, how helpful they found it, and how likely they would be to recommend it to others. Scores range from 1 to 5 for each item, where higher values represent greater satisfaction and acceptability.

SECONDARY OUTCOMES:
Values clarity | Measured at baseline and post-treatment (1 month) assessments.
  Values clarity will be measured with the Values Clarity and Awareness Interview (VCAI), an unstructured clinical interview adapted from a previous self-report measure of values clarity constructed by Forman and colleagues. The VCAI was chosen because it is the only existing measure of values clarity. Scores range from 0 to 3 for each value described, where higher values represent greater values clarity. Scores for each value described are then averaged to compute an overall clarity score.
Values awareness | Measured at baseline and post-treatment (1 month) assessments.
  Values awareness will be measured with the Values Clarity and Awareness Interview (VCAI), an unstructured clinical interview adapted from a previous self-report measure of values clarity constructed by Forman and colleagues. The VCAI was chosen because it is the only existing measure of values awareness. Scores range from 0 to 4, where higher values represent greater values awareness.
Values-congruent weight control behavior | Measured at baseline and post-treatment (1 month) assessments.
  The consistency with which individuals enact weight control behaviors in accordance with their values will be measured using an adapted Valued Living Questionnaire (VLQ) that assesses valued living as it relates to weight control in particular. Scores range from 1-10 for each of 10 valued domains of living, where higher scores represent greater personal importance and consistency with one's values.
Weight | Measured at baseline, 1 week, 2 weeks, 3 weeks, and post-treatment (1 month) assessment.
  Weight will be measured in street clothes without shoes using a lab-grade, standardized Seca® scale (accurate to 0.1 kg).
Autonomous motivation | Measured at baseline and post-treatment (1 month) assessments.
  Autonomous motivation to enact health behaviors will be measured using the Autonomous Motivation subscale of an adapted Treatment Self-Regulation Questionnaire (TSRQ) for weight loss. Scores range from 1-7, where higher scores represent greater autonomous motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Diane H Dallal, B.A., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No